CLINICAL TRIAL: NCT01108718
Title: Study of Mattress Type in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIMC 015-09
Record Dates: First submitted 2010-03-23; First posted 2010-04-22 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Fibromyalgia
Keywords: Mattress; Tempur-Pedic; Fibromyalgia; Sleep patterns
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants: Tempur Pedic first. (Experimental): Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder who receive the Tempur-Pedic mattress first, then the Control Mattress.
  Interventions: Other: Tempur-Pedic Mattress (2 months)
- Participants: Control Mattress first. (Placebo Comparator): Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the control mattress first, then the Tempur-pedic mattress.
  Interventions: Other: Control Mattress (2 months)

INTERVENTIONS:
Other: Tempur-Pedic Mattress (2 months) — Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the Tempur-Pedic mattress first, then the Control Mattress.
  Arms: Participants: Tempur Pedic first.
Other: Control Mattress (2 months) — Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the control mattress first, then the Tempur-pedic Mattress.
  Arms: Participants: Control Mattress first.

SUMMARY:
The purpose of this research study is to determine if a new mattress relieves the symptoms of fibromyalgia and improves sleep, and if this is the case, whether one type of mattress is better than the other in doing so.

DETAILED DESCRIPTION:
The various stages of sleep will be monitored via polysomnography(PSG) and scored to indicate the degree to which they reflect a normal sleep pattern. Changes in the severity of fibromyalgia symptoms will be assessed by tender point exam and study questionnaires administered at 2 month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects who fulfill the American College of Rheumatology's case definition for Fibromyalgia -- that is they have both wide spread pain and more than 10 of the 18 tender points
* 18 years of age or older
* Has to be on stable medications and followed by one physician

Exclusion Criteria:

* Subjects with the existence of an undiagnosed sleep disorder - namely obstructive sleep apnea or periodic leg movement syndrome
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Natelson, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Pain and Fatigue Study Center - Beth Israel Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Pain and Fatigue Study Center — http://www.painandfatigue.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from Principal Investigator's clinical practice at Beth Israel Medical Center in New York who fulfilled the 1990 case definition for fibromyalgia.
Pre-assignment Details: Subjects who displayed the existence of a previously undiagnosed sleep disorder were excluded from study participation.
Groups:
- Subjects Who Received the Tempur-Pedic Mattress First: Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the Tempur-Pedic mattress first, then the Control Mattress.
- Subjects Who Received the Control Mattress First: Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the control mattress first, then the Tempur-pedic mattress.
Period: Received First Intervention (2 Months)
Arm/Group | Subjects Who Received the Tempur-Pedic Mattress First | Subjects Who Received the Control Mattress First
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0
Period: Received Second Intervention (2 Months)
Arm/Group | Subjects Who Received the Tempur-Pedic Mattress First | Subjects Who Received the Control Mattress First
Started | 5 (Used control mattress was delivered to participant at crossover causing her to withdraw.) | 7
Completed | 4 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects Who Receive Tempur-Pedic Mattress First(2 Months): Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the Tempur-Pedic mattress first.
- Subjects Who Receive the Control Mattress First(2 Months): Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the control mattress first.
- Total: Total of all reporting groups
Arm/Group | Subjects Who Receive Tempur-Pedic Mattress First(2 Months) | Subjects Who Receive the Control Mattress First(2 Months) | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mattress Preference of Fibromyalgia Patients
Description: Study patients were asked to rate each test mattress after 2 months of use, based on their quality of sleep and severity of symptoms relating to fibromyalgia. The various stages of sleep were monitored via polysomnography(PSG) and scored to indicate the degree to which they reflect a normal sleep pattern. Change in severity of fibromyalgia symptoms were assessed by chi-squared and t-test.
Time Frame: 6 months
Population: Following 2 months use of each test mattress, the study patients' sleep patterns and severity of fibromyalgia symptoms were assessed. At the end of the study, study patients were asked to rate each mattress in order of preference.
Measure: Number; unit: percentage of study participants
Groups:
- All Participants: All subjects used a tempur-pedic mattress and control mattress to sleep on in a cross over design for a period of 2 months per mattress.
Arm/Group | All Participants
Number analyzed (Participants) | 11
percentage of study participants
  Tempur-Pedic Mattress | 45 [5 to 95]
  Control Mattress | 55
  No Preference | 0
Statistical Analysis 1: Comparison: All Participants; h0: Rate Preference Tempur-pedic mattress = Rate Preference control mattress h1: Rate Preference Tempur-pedic mattress = Rate Preference control mattress; Test type: Superiority or Other; p > 0.1, McNemar; Rate of Preference = .45, 95% CI 2-sided [.43 to .47], Standard Deviation .5 — Rate of preference refers specifically to Tempur-Pedic Mattress

ADVERSE EVENTS:
Groups:
- Subjects Who Received Tempur-Pedic Mattress First: Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the Tempur-Pedic mattress first.
- Subjects Who Received the Control Mattress First: Female subjects, aged 18 years or older who have been diagnosed with fibromyalgia and do not possess any sleep disorder receiving the control mattress first.
Arm/Group | Subjects Who Received Tempur-Pedic Mattress First | Subjects Who Received the Control Mattress First
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 1/5 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Who Received Tempur-Pedic Mattress First (N=5) | Subjects Who Received the Control Mattress First (N=7)
Subject's own Mattress Discarded (Investigations) | 1 (1) | 0 (0) — Subject became upset after her own mattress was mistakenly discarded during the study. Subject withdrew from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No